CLINICAL TRIAL: NCT00928655
Title: Continuous Positive Airway Pressure (CPAP) and Acetazolamide for Treatment of Patients With the Obstructive Sleep Apnea Syndrome at Altitude
Brief Title: Continuous Positive Airway Pressure and Acetazolamide to Treat Sleep Apnea Syndrome Patients at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK-1522A#1-4
Record Dates: First submitted 2009-06-22; First posted 2009-06-26 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: apnea; sleep; altitude; hypoxia; treatment; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Hypoxia | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetazolamide (Experimental): combination of acetazolamide and nocturnal continuous positive airway pressure ventilation
  Interventions: Drug: acetazolamide; Procedure: nocturnal continuous positive airway pressure
- placebo capsules (Placebo Comparator): combination of placebo and nocturnal continuous positive airway pressure ventilation
  Interventions: Procedure: nocturnal continuous positive airway pressure; Drug: placebo

INTERVENTIONS:
Drug: acetazolamide — acetazolamide 250mg 1/0/2
  Other Names: Diamox (trade name)
  Arms: acetazolamide
Procedure: nocturnal continuous positive airway pressure — continuous positive airway pressure
  Other Names: placebo capsules
Drug: placebo — placebo capsules
  Other Names: placebo capsules
  Arms: placebo capsules

SUMMARY:
The purpose of the study is to investigate the effect of nasal continuous positive airway pressure in combination with acetazolamide as a treatment for sleep related breathing disturbances in patients with the obstructive sleep apnea syndrome living at low altitude during a sojourn at moderate altitude.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome, successfully on CPAP therapy
* Residence at low altitude (< 800 m)
* Obstructive apnea/hypopnea index >20/h and a complaint of excessive daytime sleepiness before introduction of CPAP therapy
* > 15 oxygen desaturations/h (> 3% dips) during an ambulatory nocturnal pulse oximetry performed at the end of a 4-night period without CPAP

Exclusion Criteria:

* Sleep disorders other than OSA
* More than mild cardiovascular disease, unstable cardiovascular disease
* Any lung disease, pulmonary hypertension
* Chronic rhinitis
* Treatment with drugs that affect respiratory center drive (benzodiazepines or other sedatives or sleep inducing drugs, morphine or codeine derivates), stimulants (modafinil, methylphenidate, theophylline)
* Internal, neurologic or psychiatric disease that interfere with sleep quality
* Previous intolerance to moderate or low altitude (< 2600 m)
* Exposure to altitudes > 1500m for > 1 day within the last 4 weeks before the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
sleep disordered breathing and oxygenation | day 2 and 3 at altitude

SECONDARY OUTCOMES:
sleep quality, vigilance, acute mountain sickness, blood pressure | day 2 and 3 at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Director — University Hospital of Zurich, Pulmonary Division and Sleep Disorders Centre, Zurich, Switzerland
Locations (1):
- University Hospital of Zurich, Pulmonary Division and Sleep Disorders Centre, Zurich, Switzerland

REFERENCES:
- [Background] Latshang TD, Nussbaumer-Ochsner Y, Henn RM, Ulrich S, Lo Cascio CM, Ledergerber B, Kohler M, Bloch KE. Effect of acetazolamide and autoCPAP therapy on breathing disturbances among patients with obstructive sleep apnea syndrome who travel to altitude: a randomized controlled trial. JAMA. 2012 Dec 12;308(22):2390-8. doi: 10.1001/jama.2012.94847. PMID 23232895
- [Background] Latshang TD, Bloch KE, Lynm C, Livingston EH. JAMA patient page. Traveling to high altitude when you have sleep apnea. JAMA. 2012 Dec 12;308(22):2418. doi: 10.1001/jama.2012.4097. No abstract available. PMID 23232901
- [Background] Latshang TD, Bloch KE. How to treat patients with obstructive sleep apnea syndrome during an altitude sojourn. High Alt Med Biol. 2011 Winter;12(4):303-7. doi: 10.1089/ham.2011.1055. PMID 22206552
- [Background] Stadelmann K, Latshang TD, Nussbaumer-Ochsner Y, Tarokh L, Ulrich S, Kohler M, Bloch KE, Achermann P. Impact of acetazolamide and CPAP on cortical activity in obstructive sleep apnea patients. PLoS One. 2014 Apr 7;9(4):e93931. doi: 10.1371/journal.pone.0093931. eCollection 2014. PMID 24710341